CLINICAL TRIAL: NCT06263556
Title: Effectiveness of Transcutaneous Posterior Tibial Nerve Stimulation in Multiple Sclerosis Patients With Lower Urinary Track Symptoms: A Sham Controlled Prospective Randomized Controlled Study
Brief Title: Effectiveness of TTNS in MS Patients With Lower Urinary Track Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Sibel Caglar Okur, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/389
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms
Keywords: Multiple Sclerosis; Lower Urinary Track Symptoms; LUTS; Posterior tibial nerve stimulation; TPTNS; TTNS
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized and assigned to either group.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor exercises and Transcutaneous tibial nerve stimulation (Experimental): Patients in this group will receive pelvic floor exercise program as described before and transcutaneous tibial nerve stimulation (TTNS).
  The intervention will comprise 12 session of transcutaneous tibial nerve stimulation (Twice a week, for 6 continuous weeks). Each session will last 30 minutes. Two self adhesive surface electrodes will be positioned according to the protocol used by Booth et al and Sonmez et al, with the negative electrode 2 cm behind the medial malleolus, and positive electrode 10 cm proximal to it. Correct positioning will be determined by noting a hallux reaction (plantar flexion of great toe). Stimulation will be delivered at fixed frequency of 20 Hz and pulse width of 200 ms. The intensity level of the stimulation current (range 0-50 mA) will be determined once hallux reaction is observed, according to patient's tolerance.
  Interventions: Behavioral: Pelvic floor exercises; Device: Transcutaneous posterior tibial nerve stimulation
- Pelvic floor exercises and Sham Stimulation (Sham Comparator): Patients in this group will receive pelvic floor exercise program as described before and Sham stimulation.
  The intervention will comprise 12 session of sham stimulation. (Twice a week, for 6 continuous weeks) Each session will last 30 minutes. Two self adhesive surface electrodes will be positioned According to the protocol used by Booth et al, with the negative electrode 2 cm behind the lateral malleolus, and positive electrode 10 cm proximal to it, therefore avoiding the posterior tibial nerve. The stimulation current will be reduced to 2 mA once the tingling sensation is obtained and patients will be informed that they may not feel electrical sensation during the session. Stimulation will be delivered at fixed frequency of 20 Hz and pulse width of 200 ms.
  If willing, patients in this group will receive TTNS treatment after the study is completed.
  Interventions: Behavioral: Pelvic floor exercises; Device: Sham stimulation

INTERVENTIONS:
Behavioral: Pelvic floor exercises — Patients will be informed about pelvic floor muscles functions and written material will be given for home training.
  Exercise program will be planned as 1 set, 3 times per day. Each set will include 10 pelvic floor contractions. Patient will be instructed to squeeze their pelvic muscles and keep them contracted for 8 seconds. Due to fatigue and spasticity patients may experience, patients will set their own resting periods between contractions. Patients will be told to avoid contracting abdominal and gluteal muscles and avoid holding their breathe during the exercise.
  Patients will be instructed to perform exercise as following:
  1. Lie on your back. Take a deep breathe. Relax your abdominal muscles as you breathe out.
  2. Focus on your pelvic floor muscles. Squeeze your muscles as you are trying to stop the flow of your urine and stay contracted for 8 seconds, then relax.
  3. Repeat when you feel ready. You need to repeat this 10 times.
  4. Repeat this exercise 3 times per day
Device: Transcutaneous posterior tibial nerve stimulation — Patients in TTSN group will receive posterior tibial nerve stimulation based on the protocol explained before.
  Arms: Pelvic floor exercises and Transcutaneous tibial nerve stimulation
Device: Sham stimulation — Patients in sham stimulation group will receive sham stimulation based on the protocol explained before.
  Arms: Pelvic floor exercises and Sham Stimulation

SUMMARY:
Multiple sclerosis (MS) is the most common inflammatory disease of the central nervous system. It is characterized with demyelinated plaques affecting subcortical, brain stem, and spinal cord nerve fibers. During the course of the disease, with the affection myelinated nerve tracks, lower urinary track symptoms may occur. 50-90% of the MS patients experience lower urinary track symptoms (LUTS) such as urinary incontinence, urgency, nocturia and/or urinary frequency during the at one point of their life.

Aim of this study is to determine the effects of transcutaneous tibial nerve stimulation (TTNS) on symptoms and quality of life in MS patients with LUTS.

DETAILED DESCRIPTION:
This is a single-centered, prospective, single blind, randomized controlled study of patients with MS who suffer lower urinary track symptoms. All patients will be informed of the details of all the procedures and of the details of the study. After the written informed consent is obtained, patients will be distributed to two equal groups using randomized number table.

At the beginning and end of the study, post-void residue (PVR) will be calculated with ultrasonography, International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF), Incontinence Quality of Life( I-QOL), 3 day bladder diary (number of urination, urge, incontinence, nocturia) forms will be administered.

Patients will be evaluated via PVR, urodynamic measurements, ICIQ-SF, I-QOL and bladder diary.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer Adults (Age 18-50)
* Diagnosis of Multiple Sclerosis
* Expanded Disability Status Scale (EDSS) 0-6,5
* Lower urinary track symptoms (Urinary incontinence, urgency, nocturia and/or urinary frequency)
* Diagnosis of bladder disfunction with Urodynamic study within 1 months

Exclusion Criteria:

* Age less then 18
* Pacemaker or implantable defibrillator usage
* Diabetic polyuria
* Bleeding diathesis or severe bleeding tendency
* Pelvic floor disfunction or nerve damage effecting tibial nerve
* Currently pregnant or planning pregnancy
* Active urinary infection
* Active malignancy
* Severe mental disability
* Cognitive deficit
* Expanded Disability Status Scale (EDSS) greater than or equal to 7
* Unable to attend to TPTNS treatment 2 times a week
* Urodynamic findings of bladder outlet obstruction
* Surgical history because of urinary incontinence
* Urologic surgical history because of lower urinary track disfunction or symptoms
* Diagnosis of prostatic enlargement
* Diagnosis of pelvic organ prolapse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Incontinence Quality of Life (I-QOL) | 6 weeks (Before and after the treatment)
  I-QOL is used for evaluation of quality of life in patients with incontinence. It comprises 22 questions presented under three subscales: limiting behavior, psychosocial impact, and social embarrassment. All the questions are based on a five-point Likert scale (1 = a lot, 2 = quite a bit, 3 = moderate, 4 = a little, and 5 = not at all). Points obtained by each question are added together which results in a total point of 0 to 110. This total point is then recalculated to take a value between 0-100 for better understand. Higher scores indicate a better quality of life. Validation of turkish version is available.

SECONDARY OUTCOMES:
Post-void residue (PVR) | 6 weeks (Before and after the treatment)
  Post-void residue (PVR) will be calculated with ultrasonography. Evaluation will be made by same person in all patients after urination, in supine position transabdominally with 2-5 Mhz convex probe using E-Saote Mylab Seven (Italy) device.
Bladder diary | 6 weeks (Before and after the treatment)
  2 or 3 day bladder diary is recommended by European Association of Urology in patients with lower urinary track symptoms. Urination frequency, urgency, incontinence and nocturia will be evaluated using 3 day bladder diary.
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | 6 weeks (Before and after the treatment)
  ICIQ-SF allows the assessment of incontinence's severity, frequency and its impact on quality of life. ICIQ-SF scoring is also a practical and reliable method for baseline and post-treatment evaluation of patients with urge incontinence. It contains six questions. First and second questions are about demographics and the sixth question is about conditions that lead to incontinence. First, second and sixth questions have no point value. Total score varies between 0 and 21 and is obtained by adding third, fourth and fifth question's points. Higher scores indicate greater problems with incontinence. Validation of turkish version is available.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel CAGLAR, Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Arda can Kasap, Study Chair — Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kabay SC, Yucel M, Kabay S. Acute effect of posterior tibial nerve stimulation on neurogenic detrusor overactivity in patients with multiple sclerosis: urodynamic study. Urology. 2008 Apr;71(4):641-5. doi: 10.1016/j.urology.2007.11.135. PMID 18387393
- [Background] Perez DC, Chao CW, Jimenez LL, Fernandez IM, de la Llave Rincon AI. Pelvic floor muscle training adapted for urinary incontinence in multiple sclerosis: a randomized clinical trial. Int Urogynecol J. 2020 Feb;31(2):267-275. doi: 10.1007/s00192-019-03993-y. Epub 2019 Jun 10. PMID 31183535
- [Background] Celiker Tosun O, Kaya Mutlu E, Ergenoglu AM, Yeniel AO, Tosun G, Malkoc M, Askar N, Itil IM. Does pelvic floor muscle training abolish symptoms of urinary incontinence? A randomized controlled trial. Clin Rehabil. 2015 Jun;29(6):525-37. doi: 10.1177/0269215514546768. Epub 2014 Aug 20. PMID 25142280
- [Background] Booth J, Hagen S, McClurg D, Norton C, MacInnes C, Collins B, Donaldson C, Tolson D. A feasibility study of transcutaneous posterior tibial nerve stimulation for bladder and bowel dysfunction in elderly adults in residential care. J Am Med Dir Assoc. 2013 Apr;14(4):270-4. doi: 10.1016/j.jamda.2012.10.021. Epub 2012 Nov 30. PMID 23206722
- [Background] Sonmez R, Yildiz N, Alkan H. Efficacy of percutaneous and transcutaneous tibial nerve stimulation in women with idiopathic overactive bladder: A prospective randomised controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101486. doi: 10.1016/j.rehab.2021.101486. Epub 2021 Nov 11. PMID 33429090
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Cetinel B, Ozkan B, Can G. The validation study of ICIQ-SF Turkish version. Turkish J Urol 2004;30(3):332-338.
- [Background] Seckiner I, Yesilli C, Mungan NA, Aykanat A, Akduman B. Correlations between the ICIQ-SF score and urodynamic findings. Neurourol Urodyn. 2007;26(4):492-494. doi: 10.1002/nau.20389. PMID 17304520
- [Background] Wagner TH, Patrick DL, Bavendam TG, Martin ML, Buesching DP. Quality of life of persons with urinary incontinence: development of a new measure. Urology. 1996 Jan;47(1):67-71; discussion 71-2. doi: 10.1016/s0090-4295(99)80384-7. PMID 8560665
- [Background] Patrick DL, Martin ML, Bushnell DM, Yalcin I, Wagner TH, Buesching DP. Quality of life of women with urinary incontinence: further development of the incontinence quality of life instrument (I-QOL). Urology. 1999 Jan;53(1):71-6. doi: 10.1016/s0090-4295(98)00454-3. PMID 9886591
- [Background] Ozerdogan N, Beji NK, Yalcin O. Urinary incontinence: its prevalence, risk factors and effects on the quality of life of women living in a region of Turkey. Gynecol Obstet Invest. 2004;58(3):145-50. doi: 10.1159/000079422. Epub 2004 Jun 29. PMID 15237249
- [Background] Eyigor S, Karapolat H, Akkoc Y, Yesil H, Ekmekci O. Quality of life in patients with multiple sclerosis and urinary disorders: reliability and validity of Turkish-language version of Incontinence Quality of Life Scale. J Rehabil Res Dev. 2010;47(1):67-71. doi: 10.1682/jrrd.2009.08.0132. PMID 20437328
- [Background] Groen J, Pannek J, Castro Diaz D, Del Popolo G, Gross T, Hamid R, Karsenty G, Kessler TM, Schneider M, 't Hoen L, Blok B. Summary of European Association of Urology (EAU) Guidelines on Neuro-Urology. Eur Urol. 2016 Feb;69(2):324-33. doi: 10.1016/j.eururo.2015.07.071. Epub 2015 Aug 22. PMID 26304502
- [Background] Nambiar AK, Bosch R, Cruz F, Lemack GE, Thiruchelvam N, Tubaro A, Bedretdinova DA, Ambuhl D, Farag F, Lombardo R, Schneider MP, Burkhard FC. EAU Guidelines on Assessment and Nonsurgical Management of Urinary Incontinence. Eur Urol. 2018 Apr;73(4):596-609. doi: 10.1016/j.eururo.2017.12.031. Epub 2018 Feb 3. PMID 29398262
- [Background] Roehrborn CG, Peters PC. Can transabdominal ultrasound estimation of postvoiding residual (PVR) replace catheterization? Urology. 1988 May;31(5):445-9. doi: 10.1016/0090-4295(88)90746-7. PMID 3284155